CLINICAL TRIAL: NCT06715605
Title: A Controlled Phase II Clinical Trial Evaluating the Safety and Efficacy of Myelin-peptide Loaded tolDC as Treatment for Multiple Sclerosis
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of Myelin-peptide Loaded tolDC as Treatment for MS
Acronym: MS-tolDC_2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility issues, insufficient funding, delays due transition to CTIS.
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Hospital Germans Tríes i Pujol de Badalona (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCRG22-002; 2024-512891-37-00 (EU CTIS Number); 2022-003465-38 (EudraCT Number)
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: patient safety; tolerogenic dendritic cells; tolDC; phase II; MS; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intradermal arm: tolerogenic dendritic cells (tolDC) (Experimental): Each vaccine (15x106cells in 500 µL NaCl 0.9% solution supplemented with 5% human albumin) will be administered through intradermal injection at 5 sites (100 µL/site) in the posterior neck region to ensure lymphatic drainage to superficial and deep cervical lymph nodes (5-10 cm from the cervical lymph nodes). Injection sites will alternate between left and right sides
  Interventions: Biological: tolerogenic dendritic cells (tolDC)
- Control arm: standard-of-care (Active Comparator): Participants who receive standard-of-care, on first-line treatment (interferon-beta, glatiramer acetate, teriflunomide, dimethylfumarate, ponesimod, ozanimod). They will follow the same assessments as the interventional arms
  Interventions: Biological: Standard-of-care

INTERVENTIONS:
Biological: tolerogenic dendritic cells (tolDC) — In brief, clinical-grade tolDC vaccines will be prepared from leukapheresis starting material of non-mobilized blood and subsequent immunomagnetic selection of CD14+ monocytes using a CliniMACS device. CD14+ monocytes will then be cultured in GMP-grade cell culture medium supplemented with 2% human AB serum, GM-CSF, IL-4 and 1 alpha,25 dihydroxyvitamin D3. At day 4, tolDC will be stimulated using a cytokine cocktail to induce a migratory phenotype. At day 6, tolDC will be harvested, loaded with antigen, resuspended, and cryopreserved. Separate aliquots of the cell product are prepared for final quality control and quality assurance (QC/QA) assessment. This includes cell count, viability, phenotypic analysis using flow cytometry, and induction of T cell hyporesponsiveness in allo-MLR.
  Arms: Intradermal arm: tolerogenic dendritic cells (tolDC)
Biological: Standard-of-care — Standard-of-care on first-line treatment such as interferon-beta, glatiramer acetate, teriflunomide, dimethylfumarate, ponesimod and ozanimod.
  Arms: Control arm: standard-of-care

SUMMARY:
The investigators propose to design and conduct a phase II clinical trial to treat patients with multiple sclerosis (MS) by vaccination with tolerogenic dendtritic cells (tolDC), generated using Good Manufacturing Practices (GMP). Hereby, the investigators want to demonstrate the efficacy of administrating clinical-grade vitamin D3-treated tolDC loaded with myelin-derived peptides to treat a well-defined population of MS patients. In vitro generation of dedicated and stable immunomodulatory DC followed by in vitro loading of antigens to ensure tolerance and safety of DC-directed therapy is a promising strategy with the potential to induce long term tolerance

DETAILED DESCRIPTION:
A two-arm non-randomized controlled phase II clinical trial will be conducted in a coordinated and comprehensive manner to provide proof-of-concept for efficacy and safety. The primary objective of the phase II study is to determine whether tolDC-based therapy is effective and safe based on a surrogate outcome measure as primary outcome (i.e. brain MRI). Adverse events, clinical relapse rates, neurological disability (assessed using various scales) and MRI endpoints will be followed and measured over the course of 18 months. Participants who receive the tolDC treatment will be compared to MS patients, who receive standard-of-care (control group). Completion of screening assessments and confirmation of eligibility criteria should take no longer than 8 weeks. Furthermore, patients for the two arms will be recruited simultaneously and at the same pace.

ELIGIBILITY:
Inclusion Criteria:

* RIS, CIS or MS according to most recent Mc Donald's diagnostic criteria (1);
* Age 18-60 years;
* Expanded disability status scale (EDSS) of 0-6.0 inclusive;
* Active RIS, CIS, MS (relapsing and progressive forms): 1 relapse in the past year and/or at least 1 enhancing lesion on brain MRI in the past year and/or at least 1 new or enlarging T2 lesion in comparison with a reference scan from maximum 1 year before;
* RIS, CIS, MS patients already on first-line treatment or who will start first-line treatment (control arm)
* Untreated patients who do not want to be treated with currently available disease-modifying treatments or presence of treatment-related side effects; intervention arm;
* No evidence of relapse in the month prior to start of screening and throughout the screening phase;
* Only for the intervention arm: Normal total lymphocyte count above 800/mm3;
* Only for the intervention arm: Normal peripheral B cell count between 0.07x106 cells/ml and 0.53x106 cells/mL;
* Able to sign informed consent;
* Ability to comply with the protocol assessments;
* Appropriate venous access;
* Use of adequate contraceptive measures during the duration of the trial. Women and men of reproductive potential can only be included in the study following use of adequate contraceptive measures. Accepted methods of contraception include use of hormonal contraceptives (oral, intravaginal, intrauterine, or transdermal), intrauterine devices, sterilization or postmenopausal status, use of condoms with spermicide.

Exclusion Criteria:

For tolDC intradermal arm:

* Previous use of severe immunosuppressive or cytostatic treatment, including cyclophosphamide, mitoxantrone, bone marrow transplantation or (hematopoietic or mesenchymal) stem cell transplantation (at any time) prior to enrolment;
* Previous use of cladribine with last course within last 2 years or alemtuzumab with last course within last 4 years; lymphocyte counts should be above 800/mm3
* Only for the intervention arm: Use of interferon beta and glatiramer acetate in the 4 previous weeks; use of teriflunomide in the previous 4 weeks with accelerated elimination procedure; use of dimethyl/diroximel fumarate in the previous 4 weeks with normal lymphocyte counts (above 800/mm3)
* Only for the intervention arm: Treatment with fingolimod, siponimod, ponesimod, ozanimod, natalizumab, intravenous or subcutaneous immunoglobulins or plasmapheresis in the past 3 months; teriflunomide in the previous 15 weeks without accelerated elimination; anti-CD20 monoclonal antibody (including ofatumumab, rituximab and ocrelizumab) within the past 6 months prior to the first administration and until confirmation of B cell count normalization; for S1P modulators lymphocyte counts should be above 800/mm3
* Use of another investigational product in the past 6 months or longer depending on the mode of action
* Previous use of azathioprine or methotrexate in the past 3 months; lymphocyte counts should be above 800/mm3
* Previous use of other immunosuppressive agents washout is at least 3 months or longer depending on the mode of action and half-life; lymphocyte counts should be above 800/mm3

For intradermal and control arm:

* Relapse / use of corticosteroids for any reason in the previous month;
* Pregnancy or planning pregnancy in the next 18 months and breast feeding;
* Fertile patients, both men and women, who are not using an adequate method of contraception. If the patient is menopausal or sterile, it must be documented in the medical history;
* Drug or alcohol abuse;
* Inability to undergo MRI assessments or unwillingness to receive gadolinium administration;
* History of or actual signs of immunodeficiency (with the exception of treatment effects of patients on 1st line DMT) or malignancies;
* History of oncological diseases, with the exception of completely removed local basal cell carcinoma
* Concurrent clinically relevant cardiac, immunological, pulmonary, neurological, renal or other major disease;
* Positive hepatitis B or C, HIV serology, syphilis or tuberculosis indicating an active of chronic infection;
* Splenectomy;
* Dementia or severe psychiatric, cognitive or behavioral problems or other comorbidity that could interfere with the compliance to the protocol;
* Participating in another interventional clinical trial, assessing an IMP, or having participated in one, in the last 6 months.
* Previous treatment in the phase I clinical trial with tolDC.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Number of new and/or enlarging T2 lesions on MRI) | 18 months
  To evaluate the radiological efficacy of tolDC administration, number of new and/or enlarging T2 lesions on MRI scans
Safety (Occurrence and severity of adverse events will be recorded) | 18 months
  To evaluate the safety of administering tolDC, the occurrence and severity of adverse events will be recorded.

SECONDARY OUTCOMES:
Expanded disability status scale (EDSS) | 18 months
  The patients' disability level well be checked during every visit. The EDSS consists of a 10-point scale of disease severity ranging from 0, i.e. no disability, to 10, i.e. death from MS.
9 Hole Peg Test (9HPT) | 18 months
  This is a brief, standardized, quantitative test of upper extremity function
25 Foot walk test (T25FW) | 18 months
  This is a quantitative mobility and leg function performance test based on a timed 25-walk.
Symbol Digit Modalities test (SDMT) | 18 months
  This test quickly screens for organic cerebral dysfunction.
Non-clinical outcome measure (T2 lesion volume on MRI) | 18 months
  T2 lesion volume on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution in comparison to standard of care.
Non-clinical outcome measure (atrophy rate on MRI) | 18 months
  Atrophy rate on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution in comparison to standard of care.
Non-clinical outcome measure (total brain volume on MRI) | 18 months
  Total brain volume on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution in comparison to standard of care.
Non-clinical outcome measure (fractional anisotropy on MRI) | 18 months
  Fractional anisotropy on MRI scans will be evaluated to determine if administration of tolDC influences clinical and subclinical disease evolution in comparison to standard of care.

OTHER OUTCOMES:
Immunological response | 18 months
  In addition to (whole-blood) lymphocyte phenotyping and cytokine profiling before, during and after completion of the vaccination cycle, the ability of tolDC to suppress pathogenic T responses will be assessed. Therefore, myelin-specific T reactivity will be determined before, during and after completion of the vaccination cycle at specific timepoints.
Visual Analogic Scale (VAS) | 18 months
  Measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Cools, Principal Investigator — Universiteit Antwerpen; Zwi Berneman, Study Director — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Belgium